CLINICAL TRIAL: NCT06515171
Title: Efficacy and Safety of Bowel Preparation for Patency Capsule in Crohn's Disease Patients Who Previously Failed Patency Capsule
Brief Title: Efficacy and Safety of Bowel Preparation for Patency Capsule in CD Patients Who Previously Failed Patency Capsule
Status: Active, not recruiting | Type: Observational
Sponsor: Shmuel Kivity, MD (Other Government)
Responsible Party: Sponsor-Investigator, Shmuel Kivity, MD, Professor, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: 0292-19-TLV
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Crohn Disease; Crohn Disease of Small Intestine
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CD patients referred for PC before VCE: No intervention will be administered. Endoscopic capsule protocol will be performed in a uniform manner on all participants in the study as part of their routine clinical evaluation regardless of the study.
  The patient will report capsule expulsion and send a photo for documentation or report the result of the abdominal X-ray preformed 28-30 hours post swallowing
- CD patients who failed to pass an initial protocol PC on a previous attempt.: All the patients who failed the PC test will be scheduled for another test with a different preparation protocol, a common practice also today. This will be done as a standard procedure, in the clinical setting of the endoscopic capsule clinic and not as part of the study. Again, the patient will report capsule expulsion and send a photo for documentation or report the result of the abdominal X-ray preformed 28-30 hours post swallowing. If the second test was positive as well, an abdominal x-ray will be performed within 2 weeks to rule out PC retention - standard protocol for PC retention.

SUMMARY:
The goal of this observational study is to evaluate the success rate of a second bowel preparation protocol for patency capsule (PC) in Crohn Disease (CD) patients who failed to pass an initial protocol PC on a previous attempt.

The main question it aims to answer is what is the percentage of patients successfully passing the second PC test, among those who failed the first attempt.

Participants who will fail the PC test will be scheduled for another test with a different preparation protocol.

Participants will be asked to report capsule expulsion and send a photo for documentation or report the result of the abdominal X-ray preformed 28-30 hours post swallowing.

.

DETAILED DESCRIPTION:
Crohn's disease (CD) involves the entire length of the gastrointestinal tract, including a large proportion of patients with small bowel involvement. Most of the small bowel length is not accessible by conventional endoscopy for diagnosis and routine follow-up. During their lifetime these patients require repeated evaluation of disease activity and extent. Traditionally this evaluation is achieved by periodic CT or MR enterography that involves repeated exposure to radiation and contrast materials and does not provide good mucosal assessment. The use of video capsule endoscopy (VCE) among CD patients provides a good mucosal assessment without exposure to radiation or contrast material, or the risks of conventional endoscopy and sedation.

The caveat of VCE in CD is the concern of capsule retention due to strictures which are sometimes asymptomatic. This is more pronounced in patients with clinical or radiographic features implying small bowel obstruction: stricturing /fistulizing disease phenotype, abdominal pain and bloating after meals, improvement with liquid diet, stenosis and proximal dilatation on imaging studies. In these high-risk patients a patency capsule (PC) test is recommended prior to VCE. The PC is a capsule in similar dimensions to that of the VCE which contains radio-opaque components and a cellophane coat that dissolves after approximately 30 hours. Patients failing to pass the pill after 30 hours continue assessment with plain abdominal X-ray imaging or a dedicated scanner in order to confirm or deny PC expulsion. If the test is positive and the PC was not expelled, the recommendation is to avoid VCE use and limit the patient to periodical imaging and conventional endoscopy as mentioned earlier. The probability for a positive PC test is 20-30% in high risk CD patients and thus, paradoxically, some of the patients who may benefit the most from VCE, will not undergo it. Nevertheless, VCE retention rate is estimated to occur in ~ 2% of patients. However, both PC and VCE are considered safe procedures and complications even in case of capsule retention are rare.

Given that the normal transit time of the entire digestive tract is up to 72 hours, delayed expulsion of the PC (i.e. >30 hours) can simply be due to slow transit or large amount of content in the large bowel and not a small bowel obstruction. Currently there are no guidelines regarding PC preparation protocol, but It seems slow transit can probably be overcome by bowel preparation.

In the endoscopic capsule unit of the TLVMC, we implement routinely a second attempt for bowel preparation, in CD patients who fail their first attempt to pass the capsule. Studies evaluating the safety and efficacy of this protocol is lacking.

ELIGIBILITY:
Inclusion Criteria:

• Crohn Disease patients intendent to perform Capsule endoscopy .

Exclusion Criteria:

* Severe obstructive symptoms according to physician discretion
* Pregnancy
* Inability to sign informed consent
* Inability to complete the VCE procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CD patients referred for PC before VCE
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-09-11 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of second PC passaging | 3 years
  The percentage of patients successfully passing the second PC test, among those who fail the first attempt.

SECONDARY OUTCOMES:
PC retention | 3 years
  The rate of PC retention
VCE retention | 3 years
  The rate of VCE retention
Positive PC passage | 3 years
  The rate of positive PC in CD patients
Risk factors | 4 years
  Risk factors for positive PC

CONTACTS AND LOCATIONS:
Overall Officials: Nitsan Maharshak, MD, Principal Investigator — Sourasky Medical Center and Tel-Aviv University
Locations (1):
- Dep. of Gastroenterology, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No